CLINICAL TRIAL: NCT04176510
Title: Preventing Tipping Points in High Comorbidity Patients: A Lifeline From Health Coaches
Acronym: Tipping Points
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Clinical Directors Network (Network)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IHS-2017C3-8923; 8923 (Other: PCORI)
Record Dates: First submitted 2019-06-28; First posted 2019-11-25 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Comorbidity; Self-Management
Keywords: Comorbidity; Self-Management; Charlson Comorbidity Index; Health Coach

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient Centered Medical Home (PCMH) plus Health Coach (Experimental): A health coaching intervention that employs a positive affect/self-affirmation intervention to help motivate patients to succeed at implementing self-management by setting life goals, in addition to the usual care provided for patients with multiple chronic diseases by the The Patient-Centered Medical Home (PCMH).
  Interventions: Behavioral: Health Coach Intervention
- Patient Centered Medical Home (PCMH) (No Intervention): Usual care provided for patients with multiple chronic diseases by the Patient-Centered Medical Home (PCMH).

INTERVENTIONS:
Behavioral: Health Coach Intervention — A structured, manualized coaching intervention by a lay Health Coach that employs a standardized positive affect/self-affirmation intervention, not tied to specific chronic diseases, to help motivate patients to learn to implement self-management by setting life goals.
  Arms: Patient Centered Medical Home (PCMH) plus Health Coach

SUMMARY:
This pragmatic cluster randomized clinical trial (cRCT) aims to evaluate the comparative effectiveness (CER) of two approaches to preventing destabilization ("tipping points") that lead to unplanned hospitalization and increased disability. The cRCT compares the outcomes of patients randomized in clusters by site within four Federally Qualified Health Center (FQHC) networks in New York City (NYC) and Chicago to either: 1) the Patient Centered Medical Home (PCMH); or 2) the Patient Centered Home plus a health coaching intervention that employs a positive affect/self-affirmation intervention to help motivate patients to succeed at implementing self-management by setting life goals (experimental).

This RCT embeds novel effective interventions within large FQHC networks, namely, Community Healthcare Network and the Family Health Centers of New York University (NYU) Langone in NYC and Erie Family Health Centers and Friend Family Health Center in Chicago, serving patients with multiple chronic diseases or high comorbidity. This CER study compares two PCMH-based strategies and will provide a manualized training system that can be disseminated and implemented across the national FQHC networks, with over 9,000 delivery sites that serve nearly 25 million low-income and minority patients, and can be implemented in a wider range of practice settings, organization types and population characteristics.

Among 1920 adult patients with a Charlson Comorbidity Index ≥4 who are established primary care patients of 16 Federally Qualified Health Centers (FQHCs) in NYC (8 FQHCs) and Chicago (8 FQHCs) this pragmatic cRCT aims to evaluate the effectiveness of two approaches to preventing destabilization that leads to unplanned hospitalization and increased disability.

This Patient-Centered Outcomes Research Institute (PCORI) study builds on the National Patient-Centered Clinical Research Network (PCORnet) Clinical Data Research Networks (CDRNs) in NYC and Chicago. Patients will be identified via electronic health records (EHRs) and their outcomes assessed through comprehensive, longitudinal, electronic health records that are aggregated by these PCORnet CDRNs.

ELIGIBILITY:
Inclusion Criteria:

* Established patients of the participating Federally Qualified Health Centers (FHQCs)
* Charlson comorbidity index ≥4

Exclusion Criteria:

* Metastatic cancer,
* End stage renal disease on dialysis
* Post-transplant
* Severe mental illness
* Drug/alcohol abuse
* Cannot communicate in English or Spanish.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1920 (Estimated)
Dates: Start 2019-11-20 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of Unplanned Hospitalizations | 24 months
  Unplanned hospitalizations are hospitalizations for any reason other than elective procedures. This specifically excludes admissions for a planned procedure (i.e. elective surgery, chemotherapy, childbirth, etc.). Admissions not accompanied by an acute diagnosis are not counted. Circumstances surrounding hospitalization will be recorded through a vignette, classified by two independent blinded reviewers.
World Health Organization Disability Assessment Scale (WHODAS) Scale | 24 months
  The WHODAS 2.0 (36 items) assesses individual level of function in six major life domains: cognition (understanding and communication) mobility (move and get around), self-care (attend to personal hygiene, dress, eat and live alone), getting along (interact with other people); life activities (carry out responsibility of home, work, school), and participation in society (engage in community, civil and recreational activities).Chronbach's α was >0.79 for each of the domains. The test-retest reliability ranged from 0.93 to 0.96 at the domain level. WHODAS 2.0 generates one global score and six domain-specific scores, validated against the Short Form 36 (SF-36) Health Survey and other scales and is responsive to change.

SECONDARY OUTCOMES:
Number of Emergency Department Visits | 24 months
  This includes visits to emergency departments as captured by Encounter Type, Provider and Facility Location in Electronic Health Records.
Health Education Impact Questionnaire | 24 months
  The Health Education Impact Questionnaire evaluates eight domains: positive and active engagement in life, health directed behavior, skill and technique acquisition, constructive attitudes and approaches, self-monitoring and insight, health services navigation, social integration and support, and emotional wellbeing. Each domain is scored separately and domain scores range between 1 and 4. For the domain of emotional wellbeing, lower score represents better outcome. For all other domains, higher scores represent better outcomes.
Patient Activation Measure | 24 months
  The Patient Activation Measure (PAM-13) assesses skill and confidence for self-management of chronic conditions. It is a 13 item scale with a 5-point Likert response scale (disagree strongly, disagree, agree, agree strongly, or N/A). Raw scores are transformed to a scale of 0-100 with 100 being the highest activation and 0 the lowest activation in self-management.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan N Tobin, PhD, Principal Investigator — Clinical Directors Network; Mary Charlson, MD, Principal Investigator — Weill Medical College of Cornell University; Andrea Cassells, MPH, Study Director — Clinical Directors Network; Anisa Mian, MPH, Study Director — Clinical Directors Network
Locations (4):
- United States (4):
  - Friend Health, Inc., Chicago, Illinois
  - Erie Family Health Centers, Chicago, Illinois
  - Family Health Centers at NYU Langone, Brooklyn, New York
  - Community Healthcare Network, New York, New York

REFERENCES:
- [Derived] Charlson ME, Mittleman I, Ramos R, Cassells A, Lin TJ, Eggleston A, Wells MT, Hollenberg J, Pirraglia P, Winston G, Tobin JN. Preventing "tipping points" in high comorbidity patients: A lifeline from health coaches - rationale, design and methods. Contemp Clin Trials. 2025 May;152:107865. doi: 10.1016/j.cct.2025.107865. Epub 2025 Feb 28. PMID 40024364